CLINICAL TRIAL: NCT01871090
Title: Remote Device Interrogation In The Emergency Department
Acronym: REMEDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 60047158
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Heart Disease; Cardiovascular Disease; Heart Failure; Arrhythmias, Cardiac
Keywords: Remote Monitoring; Remote Care; Cardiac Resynchronization Therapy; Pacemaker; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interrogation with unpaired remote transmitter (Active Comparator): Interrogation with an unpaired remote monitoring transmitter for devices that are compatible.
  Interventions: Device: Unpaired remote monitoring transmitter
- Interrogation with programmer (No Intervention): Interrogation with programmer according to usual standard of care

INTERVENTIONS:
Device: Unpaired remote monitoring transmitter — Unpaired remote monitoring transmitter
  Other Names: St. Jude Medical Merlin@home remote monitoring transmitter
  Arms: Interrogation with unpaired remote transmitter

SUMMARY:
A prospective, post market, non-randomized study to evaluate the reduction in time to interrogation for patients with St. Jude Medical remote care compatible devices interrogated by the unpaired Merlin@home transmitter in the Emergency Department (ED). Two sites will enroll up to 100 patients total.

Expected duration of the study is 6 months. Once enrolled the patient will participate in the study for the duration of the Emergency Department stay, until discharged or admitted to the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Present to Emergency Department with an implanted pacemaker or defibrillator.
2. Are 18 years of age or older, or of legal age to give informed consent specific to state law.
3. Are willing and able to provide informed consent for study participation.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Girsky, MD, Principal Investigator — Los Angeles Biomedical Research Institute at Harbor - UCLA
Locations (1):
- Genesis Healthcare System, Zanesville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled from 20-September-2013 to 14-April-2015 from the Genesis Healthcare Emergency Department located in Zanesville, Ohio.
Pre-assignment Details: There were 16 screen failures because at the time of their enrollment, the patient group had met maximum enrollment for their patient group (compatible vs. non-compatible cardiac device) under the initial protocol.
Groups:
- Interrogation With Unpaired Remote Monitoring Transmitter: Interrogation with an unpaired remote monitoring transmitter for devices that are compatible.
  Unpaired remote monitoring transmitter
Period: Overall Study
Arm/Group | Interrogation With Unpaired Remote Monitoring Transmitter | Interrogation With Programmer
Started | 35 | 48
Completed | 33 | 25
Not Completed | 2 | 23
Not completed — Interrogation not done in Emergency Room | 1 | 22
Not completed — Interrogation not completed correctly | 1 | 0
Not completed — Subject Non-Compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interrogation With Unpaired Remote Monitoring Transmitter | Interrogation With Programmer | Total
Number analyzed (Participants) | 35 | 48 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (18.6) | 64.4 (14.7) | 65.5 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 7 | 24
  Male | 18 | 41 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 33 | 41 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Interrogation
Description: Time to interrogation is defined as the time from Triage (decision to interrogate the device) until the first of: Completion of interrogation, Time of Clinical/Treatment decision, or Emergency Department check out time.
Time Frame: On day of Emergency Department admission
Measure: Median (Full Range); unit: Minutes
Arm/Group | Interrogation With Unpaired Remote Monitoring Transmitter | Interrogation With Programmer
Number analyzed (Participants) | 35 | 48
Minutes | 25 [1 to 95] | 210 [1 to 980]

2. Secondary Outcome: Time to Clinical/Treatment Decision
Description: Defined as the time from the Emergency Department Check In Time until the first of: Time of Clinical/Treatment Decision or Emergency Department Check Out Time (discharged/leaves Emergency Department or admitted to hospital).
Time Frame: On day of Emergency Department admission
Measure: Median (Full Range); unit: Minutes
Arm/Group | Interrogation With Unpaired Remote Monitoring Transmitter | Interrogation With Programmer
Number analyzed (Participants) | 35 | 48
Minutes | 204 [67 to 354] | 270 [24 to 874]

3. Other Pre Specified Outcome: Length of Emergency Department Stay
Description: Defined as the time from the Emergency Department Check In Time until the Emergency Department Check Out Time (discharged/leaves Emergency Department or admitted to hospital).
Time Frame: On day of Emergency Department admission
Measure: Median (Full Range); unit: Minutes
Arm/Group | Interrogation With Unpaired Remote Monitoring Transmitter | Interrogation With Programmer
Number analyzed (Participants) | 35 | 48
Minutes | 261 [109 to 547] | 245 [66 to 874]

ADVERSE EVENTS:
Time Frame: Adverse Events were reported while subject was in the Emergency Department.
Arm/Group | Interrogation With Unpaired Remote Monitoring Transmitter | Interrogation With Programmer
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/48
Other Adverse Events (participants affected / at risk) | 1/35 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interrogation With Unpaired Remote Monitoring Transmitter (N=35) | Interrogation With Programmer (N=48)
Failed transmission from the study device to fax, email, or Merlin.Net (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
23 subjects in the control group and 2 in the study group were not included due to their interrogation not being done in the emergency department.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No